CLINICAL TRIAL: NCT03087773
Title: Impact of EMpagliflozin on Cardiac Function and Biomarkers of Heart Failure in Patients With Acute MYocardial Infarction
Acronym: EMMY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: United Arab Emirates University (Other); Medical University of Vienna (Other); Landeskrankenhaus Feldkirch (Other); Paracelsus Medical University (Other); Hospital Rudolfstiftung (Other); Klinikum Klagenfurt am Wörthersee (Other); Barmherzige Brüder Eisenstadt (Other); Cardinal Schwarzenberg Hospital (Other); Johannes Kepler University of Linz (Other); Landesklinikum Sankt Polten (Other); Landeskrankenhaus II Graz West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-2017-01
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acute Myocardial Infarction
Keywords: Biomarker; Heart failure; SGLT-2 inhibitor; Empagliflozin; Randomized controlled trial
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): The subjects will receive Empagliflozin 10mg.
  Interventions: Drug: Empagliflozin 10 mg
- Placebo Oral Tablet (Placebo Comparator): The subjects will receive placebo.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 mg — The subject will receive Empagliflozin 10 mg orally once daily for 26 weeks.
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo Oral Tablet — The subject will receive Placebo orally once daily for 26 weeks.
  Other Names: Sugar pill
  Arms: Placebo Oral Tablet

SUMMARY:
This study is planned to investigate the impact of Empagliflozin on biomarkers of heart failure in patients with myocardial infarction with and without type 2 diabetes mellitus within 6 months after the event.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is associated with an about two to three-fold increased risk for cardiovascular events as compared to subjects without diabetes.

Sodium-dependent glucose cotransporter 2 (SGLT-2) is mainly expressed in human kidneys and small intestinal cells. In the proximal tubule of the nephron SGLT-2 is responsible for the reabsorption of approximately 90% of the filtrated glucose. Inhibition of SGLT-2 was shown to increase renal glucose excretion and to lower glucose. Subsequently, a number of SGLT-2 inhibitors were developed and are currently approved for the treatment of type 2 diabetes.

Recently, Zinman et al published the results of the Cardiovascular Outcome Event Trial in Type 2 Diabetes Mellitus Patient trial (EMPA REG OUTCOME TRIAL) where the cardiovascular impact of a glucose lowering regimen including Empagliflozin as compared to usual glucose control without an SGLT-2 inhibitor was investigated. The trial demonstrated an unexpected reduction in the primary composite endpoint, comprising cardiovascular death, non-fatal myocardial infarction and non-fatal stroke. The reduction was mainly driven by a 38% relative risk reduction in cardiovascular deaths; moreover they demonstrated an impressive 35% relative risk reduction in the secondary endpoint hospitalization for heart failure. Of note, the beneficial effects observed in the Empagliflozin group seem to occur very rapidly after commencing the treatment, as suggested by the early separation of the Kaplan-Meier curves. However, the mechanisms responsible for this finding remain unclear. Diuretic effects with subsequent impact on hemodynamics or potential cardioprotective effects of glucagon, which levels rise under the treatment with SGLT-2 inhibitors and the resulting rise in ketone bodies or a small increase in hematocrit have been suggested.

The aim of our trial is to investigate whether Empagliflozin treatment commenced within 72-h after acute myocardial infarction has an impact on heart failure in subjects with and without diabetes mellitus type 2.

ELIGIBILITY:
Inclusion Criteria:

1. Myocardial infarction with evidence of significant myocardial necrosis defined as a rise in creatinine kinase >800 U/l and a troponin T-level (or troponin I-level) >10x upper limit of normal (ULN). In addition at least 1 of the following criteria must be the met:

   * Symptoms of ischemia
   * ECG (electrocardiogram) changes indicative of new ischemia (new ST-T changes or new LBBB)
   * Imaging evidence of new regional wall motion abnormality
2. 18 - 80 years of age
3. Informed consent has to be given in written form
4. estimated glomerular filtration rate (eGFR) > 45 ml/min/1.73m2
5. Blood pressure before first drug dosing: Riva Rocci (RR) systolic >110 mmHg
6. Blood pressure before first drug dosing: Riva Rocci (RR) diastolic >70 mmHg
7. ≤72h after myocardial infarction (after the performance of a coronary angiography)

Exclusion Criteria:

1. Any other form of diabetes mellitus than type 2 diabetes mellitus, history of diabetic ketoacidosis
2. Blood potential hydrogen (pH) < 7,32
3. Known allergy to SGLT-2 inhibitors
4. Hemodynamic instability as defined by intravenous administration of catecholamine, calcium sensitizers or phosphodiesterase inhibitors
5. >1 episode of severe hypoglycemia within the last 6 months and treatment with insulin or sulfonylurea
6. Females of childbearing potential without adequate contraceptive methods (i.e. sterilization, intrauterine device, vasectomized partner; or medical history of hysterectomy)
7. Acute symptomatic urinary tract infection (UTI) or genital infection
8. Patients currently being treated with any SGLT-2 inhibitor or having received treatment with any SGLT-2 inhibitor within the 4 weeks prior to the screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, Assoc.-Prof., Study Director — Medical University of Graz; Dirk von Lewinski, Assoc.-Prof., Principal Investigator — Medical University of Graz
Locations (11):
- Austria (11):
  - Barmherzige Brüder Eisenstadt, Eisenstadt, Burgenland
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Kardinal schwarzenberg Klinikum Schwarzach, Schwarzach im Pongau, Salzburg
  - Kepler Universitätsklinikum Linz, Linz, Upper Austria
  - VIVIT Institut am akademischen Lehrkrankenhaus Feldkirch, Feldkirch, Vorarlberg
  - Landeskrankenhaus Graz II Standort West, Graz
  - Medical University of Graz, Graz
  - Uniklinikum Salzburg, Salzburg
  - Krankenanstalt Rudolfstiftung, Vienna
  - Allgemeines Krankenhaus Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tripolt NJ, Kolesnik E, Pferschy PN, Verheyen N, Ablasser K, Sailer S, Alber H, Berger R, Kaulfersch C, Leitner K, Lichtenauer M, Mader A, Moertl D, Oulhaj A, Reiter C, Rieder T, Saely CH, Siller-Matula J, Weidinger F, Zechner PM, von Lewinski D, Sourij H; EMMY study group. Impact of EMpagliflozin on cardiac function and biomarkers of heart failure in patients with acute MYocardial infarction-The EMMY trial. Am Heart J. 2020 Mar;221:39-47. doi: 10.1016/j.ahj.2019.12.004. Epub 2019 Dec 12. PMID 31901799
- [Result] von Lewinski D, Kolesnik E, Tripolt NJ, Pferschy PN, Benedikt M, Wallner M, Alber H, Berger R, Lichtenauer M, Saely CH, Moertl D, Auersperg P, Reiter C, Rieder T, Siller-Matula JM, Gager GM, Hasun M, Weidinger F, Pieber TR, Zechner PM, Herrmann M, Zirlik A, Holman RR, Oulhaj A, Sourij H. Empagliflozin in acute myocardial infarction: the EMMY trial. Eur Heart J. 2022 Nov 1;43(41):4421-4432. doi: 10.1093/eurheartj/ehac494. PMID 36036746
- [Result] Benedikt M, Mangge H, Aziz F, Curcic P, Pailer S, Herrmann M, Kolesnik E, Tripolt NJ, Pferschy PN, Wallner M, Zirlik A, Sourij H, von Lewinski D. Impact of the SGLT2-inhibitor empagliflozin on inflammatory biomarkers after acute myocardial infarction - a post-hoc analysis of the EMMY trial. Cardiovasc Diabetol. 2023 Jul 5;22(1):166. doi: 10.1186/s12933-023-01904-6. PMID 37407956
- [Result] Aziz F, Tripolt NJ, Pferschy PN, Kolesnik E, Mangge H, Curcic P, Hermann M, Meinitzer A, von Lewinski D, Sourij H; EMMY Investigators. Alterations in trimethylamine-N-oxide in response to Empagliflozin therapy: a secondary analysis of the EMMY trial. Cardiovasc Diabetol. 2023 Jul 20;22(1):184. doi: 10.1186/s12933-023-01920-6. PMID 37475009
- [Result] von Lewinski D, Kolesnik E, Aziz F, Benedikt M, Tripolt NJ, Wallner M, Pferschy PN, von Lewinski F, Schwegel N, Holman RR, Oulhaj A, Moertl D, Siller-Matula J, Sourij H. Timing of SGLT2i initiation after acute myocardial infarction. Cardiovasc Diabetol. 2023 Sep 30;22(1):269. doi: 10.1186/s12933-023-02000-5. PMID 37777743
- [Result] Sourij C, Oulhaj A, Aziz F, Tripolt NJ, Aberer F, Pferschy PN, Postula M, Drexel H, Benedikt M, Kolesnik E, Pieber TR, Bugger H, von Lewinski D, Sourij H. Impact of glycaemic status on the cardiac effects of empagliflozin when initiated immediately after myocardial infarction: A post-hoc analysis of the EMMY trial. Diabetes Obes Metab. 2024 May;26(5):1971-1975. doi: 10.1111/dom.15477. Epub 2024 Jan 29. No abstract available. PMID 38287198
- [Result] Sourij C, Aziz F, Tripolt NJ, Siller-Matula J, Pferschy PN, Kolesnik E, Wallner M, Eyileten C, Postula M, Oulhaj A, Sourij H, von Lewinski D; EMMY study group. Effects of empagliflozin in women and men with acute myocardial infarction: An analysis from the EMMY trial. Hellenic J Cardiol. 2024 Jan-Feb;75:3-8. doi: 10.1016/j.hjc.2023.05.007. Epub 2023 May 24. PMID 37236318
- [Derived] Schwegel N, Strohhofer C, Kolesnik E, Oltean S, Huttmair A, Pipp C, Benedikt M, Verheyen N, Gollmer J, Ablasser K, Wallner M, Santner V, Tripolt N, Pferschy P, Zechner P, Alber H, Siller-Matula JM, Kopp K, Zirlik A, Aziz F, Sourij H, von Lewinski D. Impact of empagliflozin on cardiac structure and function assessed by echocardiography after myocardial infarction: a post-hoc sub-analysis of the emmy trial. Clin Res Cardiol. 2025 May;114(5):629-639. doi: 10.1007/s00392-024-02523-1. Epub 2024 Sep 16. PMID 39297940
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between May 2017 (FPFV) and Oct 2021 (LPFV), at 11 sites: 1) University Hospital Graz; 2) Hospital Klagenfurt 3) Brothers of Saint John of God Eisenstadt; 4) Paracelsus Medical Private University Salzburg; 5) Vorarlberg Institute for Vascular Investigation and Treatment; 6) Kardinal Schwarzenberg Hospital Schwarzach; 7) J. Kepler University Hospital Linz; 8) University Hospital St. Pölten; 9) Allgemeines Krankenhaus Vienna; 10) Hospital Graz II: 11) Hospital Landstrasse Vienna
Period: Overall Study
Arm/Group | Empagliflozin | Placebo Oral Tablet
Started | 237 | 239
Completed | 217 | 227
Not Completed | 20 | 12
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Lost to Follow-up | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | Placebo Oral Tablet | Total
Number analyzed (Participants) | 237 | 239 | 476
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [52 to 64] | 57 [52 to 65] | 57 [52 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 195 | 197 | 392
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 237 | 239 | 476
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m²] | 27.7 [25.3 to 30.3] | 27.2 [24.9 to 30.2] | 27.6 [25.1 to 30.3]
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 125 [116 to 131] | 125 [118 to 131] | 125 [117 to 131]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 78 [74 to 85] | 78 [75 to 85] | 78 [74 to 85]
Obesity [Count of Participants; unit: Participants] | 68 | 70 | 138
Type 2 diabetes [Count of Participants; unit: Participants] | 30 | 33 | 63
Hypertension [Count of Participants; unit: Participants] | 92 | 107 | 199
Dyslipidaemia [Count of Participants; unit: Participants] | 71 | 64 | 135
Smoking active or former [Count of Participants; unit: Participants] | 171 | 170 | 341
Coronary artery disease [Count of Participants; unit: Participants] | 28 | 25 | 53
History of stroke [Count of Participants; unit: Participants] | 5 | 1 | 6
History of coronary artery bypass graft [Count of Participants; unit: Participants] | 1 | 1 | 2
History of myocardial infarction [Count of Participants; unit: Participants] | 14 | 9 | 23
Depression [Count of Participants; unit: Participants] | 15 | 9 | 24
History of carcinoma [Count of Participants; unit: Participants] | 11 | 13 | 24
Coronary 3-vessel disease [Count of Participants; unit: Participants] | 50 | 36 | 86
Coronary 2-vessel disease [Count of Participants; unit: Participants] | 82 | 80 | 162
Coronary 1-vessel disease [Count of Participants; unit: Participants] | 105 | 123 | 228
Angiotensin-converting enzyme inhibitor/angiotensin receptor blocker [Count of Participants; unit: Participants] | 96 | 97 | 193
Angiotensin receptor-neprilysin inhibitor [Count of Participants; unit: Participants] | 2 | 7 | 9
Beta-blocker [Count of Participants; unit: Participants] | 223 | 234 | 457
Mineralcorticoid receptor antagonist [Count of Participants; unit: Participants] | 86 | 94 | 180
Loop diuretic [Count of Participants; unit: Participants] | 27 | 24 | 51
Statin [Count of Participants; unit: Participants] | 229 | 233 | 462
Ezetimibe [Count of Participants; unit: Participants] | 29 | 30 | 59
Calcium channel blocker [Count of Participants; unit: Participants] | 9 | 12 | 21
Aspirin [Count of Participants; unit: Participants] | 235 | 239 | 474
Anticoagulatoin drugs [Count of Participants; unit: Participants] | 16 | 21 | 37
Metformin [Count of Participants; unit: Participants] | 21 | 20 | 41
Dipeptidyl peptidase 4 inhibitor [Count of Participants; unit: Participants] | 7 | 6 | 13
Sulfonylurea [Count of Participants; unit: Participants] | 2 | 2 | 4
Glucagon-like peptide-1 receptor agonist [Count of Participants; unit: Participants] | 2 | 2 | 4
Insulin [Count of Participants; unit: Participants] | 5 | 6 | 11
N-terminal prohormone of brain natriuretic peptide [Median (Inter-Quartile Range); unit: pg/mL] | 1,272 [773 to 2,247] | 1,373 [754 to 2,217] | 1,294 [757 to 2,246]
Estimated glomerular filtration rate [Median (Inter-Quartile Range); unit: ml/min/1.73m²] | 92 [78 to 101] | 91 [78 to 102] | 92 [78 to 102]
HbA1c [Median (Inter-Quartile Range); unit: percentage of HbA1c] | 5.6 [5.4 to 6.0] | 5.7 [5.4 to 6.0] | 5.6 [5.4 to 6.0]
Creatine kinase [Median (Inter-Quartile Range); unit: U/L] | 1,668 [1,136 to 2,532] | 1,701 [1,254 to 2,404] | 1,673 [1,202 to 2,456]
Troponin T [Median (Inter-Quartile Range); unit: ng/L] | 3,059 [2,082 to 4,775] | 3,029 [1,980 to 4,856] | 3,039 [2,037 to 4,856]
Total cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 188 [163 to 225] | 188 [162 to 220] | 188 [162 to 223]
Low-density lipoprotein [Median (Inter-Quartile Range); unit: mg/dL] | 118 [96 to 150] | 121 [90 to 145] | 120 [93 to 149]
High-density lipoprotein [Median (Inter-Quartile Range); unit: mg/dL] | 44 [36 to 52] | 43 [36 to 54] | 44 [36 to 54]
Aspartate aminotransferase [Median (Inter-Quartile Range); unit: U/L] | 203 [136 to 328] | 212 [120 to 320] | 204 [125 to 322]
Alanine aminotransferase [Median (Inter-Quartile Range); unit: U/L] | 50 [37 to 75] | 50 [38 to 68] | 50 [37 to 72]
Gamma glutamyltransferase [Median (Inter-Quartile Range); unit: U/L] | 29 [21 to 49] | 32 [21 to 48] | 31 [21 to 49]

OUTCOME MEASURES:

1. Primary Outcome: Changes of Nt-proBNP (N-terminales Pro Brain Natriuretic Peptide) Levels
Description: Difference in the change of nt-proBNP (N terminales pro brain natriuretic peptide) levels between treatment groups from randomization to week 26
Time Frame: 26 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Empagliflozin | Placebo Oral Tablet
Number analyzed (Participants) | 217 | 227
pg/mL | -84.9 [-91.7 to -72.6] | -82.2 [-89.2 to -69.8]

2. Secondary Outcome: Changes in Ejection Fraction
Description: Difference in the change of ejection fraction between treatment groups from randomization to week 26 Ejection fraction was measured by ultrasound.
Time Frame: 26 weeks
Population: Total ultrasound measurements were just available from 212 (empagliflozin group) and 209 patients (placebo group).
Measure: Median (Inter-Quartile Range); unit: percentage of ejection fraction
Arm/Group | Empagliflozin | Placebo Oral Tablet
Number analyzed (Participants) | 212 | 209
percentage of ejection fraction | 4.7 [3.6 to 5.8] | 2.8 [1.8 to 3.9]

3. Secondary Outcome: Changes in Left Ventricular End-diastolic Volume
Description: Difference in the change of left ventricular end-diastolic volume from randomization to week 26 (measured by ultrasound)
Time Frame: 26 weeks
Population: Total ultrasound measurements were just available from 212 (empagliflozin group) and 209 patients (placebo group).
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Empagliflozin | Placebo Oral Tablet
Number analyzed (Participants) | 212 | 209
ml | 3.4 [-0.7 to 7.4] | 13.5 [8.7 to 18.3]

4. Secondary Outcome: Duration of Hospital Stay
Description: Difference in the duration of hospital stay between the treatment groups after initiation of the study treatment.
  This outcome measure includes all days of an inpatient stay in a hospital after the initial discharge.
Time Frame: 30 weeks
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Empagliflozin | Placebo Oral Tablet
Number analyzed (Participants) | 217 | 227
days | 6.0 [3 to 9] | 6.0 [3 to 9]

5. Secondary Outcome: Changes in E/è Ratio From Baseline to Week 26
Description: E/E' ratio is a measure of left ventricular filling pressure. The E/e' ratio is a parameter for diastolic function assessment that is frequently used for Heart failure with preserved ejection fraction evaluation.
  To derive the E/e´ ratio one must divide the maximum velocity of the E-wave of mitral valve inflow by the maximal velocity of E. In normal individuals the E/e´ ratio is <8. In the presence of diastolic dysfunction / impaired relaxation, e´ will be rather low. In contrast, the E-wave increases with elevated filling pressures. Thus the E/e´ ratio will increase in the presence of diastolic dysfunction. An E/e´ratio >14 is highly suggestive of elevated filling pressures.
Time Frame: From Baseline to Week 26
Population: Total ultrasound measurements were just available from 212 (empagliflozin group) and 209 patients (placebo group).
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Empagliflozin | Placebo Oral Tablet
Number analyzed (Participants) | 212 | 209
Ratio | -9.7 [-13.1 to -6.4] | -0.7 [-1.1 to -0.4]

6. Secondary Outcome: Changes in Left Ventricular End-systolic Volume (LVESV) From Baselin to Week 26
Description: End-systolic volume (ESV) is the volume of blood in a ventricle at the end of contraction, or systole, and the beginning of filling, or diastole.
  Left ventricular end-systolic volume (LVESV) was measured at baseline and after 26 weeks by echocardiography.
Time Frame: Baseline to Week 26
Population: Total ultrasound measurements were just available from 212 (empagliflozin group) and 209 patients (placebo group).
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Empagliflozin | Placebo Oral Tablet
Number analyzed (Participants) | 212 | 209
ml | -3.6 [-6.3 to -1.0] | 4.3 [1.2 to 7.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to visit 5 (4 weeks after the end of intervention) - in total for 30 weeks.
Description: Adverse events (AE) that occured during this study were recorded on AE case report forms. The Sponsor reported all serious AEs (SAEs) and AEs which were relevant for a reported SAE as well as Adverse Events of Special Interest by fax using Böhringer Ingelheim (BI) SAE form to the BI Unique Entry Point. The sponsor reported the SAEs to the ethics committee and the local authorities as well as Boehringer Ingelheim Pharmacovigilance in accordance with the reporting instructions.
Arm/Group | Empagliflozin | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 3/237 | 0/239
Serious Adverse Events (participants affected / at risk) | 31/237 | 32/239
Other Adverse Events (participants affected / at risk) | 18/237 | 9/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=237) | Placebo Oral Tablet (N=239)
Any hospitalisation (Cardiac disorders) | 31 (35) | 32 (34) — Empagliflozin 35 events / Placebo 34 events
Hospitalisation due to heart failure (Cardiac disorders) | 3 (6) | 4 (4) — Empagliflozin 6 events / Placebo 4 events
Hospitalisation due to cardiovascular event (Cardiac disorders) | 2 (2) | 5 (5) — Empagliflozin 2 events / Placebo 5 events
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=237) | Placebo Oral Tablet (N=239)
Urinary tract infection (Infections and infestations) | 11 (18) | 7 (8) — Empagliflozin 18 events / Plazebo 8 events
Genital fungal infection (Infections and infestations) | 7 (7) | 2 (2) — Empagliflozin 7 events / Placebo 2 events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT03087773/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT03087773/SAP_001.pdf